CLINICAL TRIAL: NCT05044468
Title: A Randomized Blinded Controlled Trial of EXPAREL vs 1% Lidocane as Local Anesthetic in Patients Undergoing Pleuroscopy With Pleural Biopsy and Indwelling Pleural Catheter Placement
Brief Title: EXPAREL or Lidocane as Local Anesthetic in Patients Undergoing Pleuroscopy With Pleural Biopsy and Indwelling Pleural Catheter Placement
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-0237; NCI-2021-08954 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0237 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-02; First posted 2021-09-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Malignant Pleural Neoplasm
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (liposomal bupivacaine) (Experimental): Patients receive liposomal bupivacaine via injection into the intercostal nerve block.
  Interventions: Drug: Liposomal Bupivacaine; Other: Questionnaire Administration
- Group B (lidocaine) (Active Comparator): Patients receive lidocaine via injection into the pleuroscopy port incision sites and indwelling pleural catheter site.
  Interventions: Drug: Lidocaine; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Lidocaine — Given via injection
  Other Names: .omega.-Diethylamino-2,6-dimethylacetanilide; 2-(Diethylamino)-2'',6''-acetoxylidide; Cuivasil; Duncaine; Leostesin; Lidothesin; Lignocaine; Rucaina
  Arms: Group B (lidocaine)
Drug: Liposomal Bupivacaine — Given via injection
  Other Names: Bupivacaine Liposome Injectable Suspension; Exparel
  Arms: Group A (liposomal bupivacaine)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial investigates the effect of EXPAREL compared to lidocane as a local anesthetic in patients who are undergoing pleuroscopy with pleural biopsy and indwelling pleural catheter placement. This trial aims to see whether EXPAREL or lidocane is able to make patients more comfortable.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare Global chest pain score (measured on the Visual Analog Scale [VAS] scale) post-procedure and post procedural chest pain (measured on the numerical rating scale), at the time of discharge from recovery between liposomal bupivacaine (EXPAREL) and 1 percent lidocaine.

SECONDARY OBJECTIVES:

I. To compare post procedural chest pain (measured on the numerical rating scale) at the time of discharge from recovery, 24 hours and 48 hours post procedure between EXPAREL and 1 percent lidocaine.

II. To assess the change in global chest pain score (measured on the VAS scale) from baseline to the time of discharge from recovery, and post procedural chest pain (measured on the numerical rating scale) from baseline over time between EXPAREL and 1 percent lidocaine.

III. To compare the number of narcotics within 24 hours, and from 24 to 48 hours post procedure between EXPAREL and 1 percent lidocaine.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP A: Patients receive liposomal bupivacaine via injection into the intercostal nerve block.

GROUP B: Patients receive lidocaine via injection into the pleuroscopy port incision sites and indwelling pleural catheter site.

ELIGIBILITY:
Inclusion criteria:

1. Referral to pulmonary services for pleuroscopy with biopsies and IPC placement/chest tube placement
2. Age > 18

Exclusion criteria:

1. Inability to provide informed consent
2. Study subject has any disease or condition that interferes with safe completion of the study including:

   a. Allergic reaction to EXPAREL
3. Need for pleurodesis
4. Allergies to lidocaine or other local anesthetics.
5. Pregnancy
6. Advanced liver disease where the clinician deems the procedure unsafe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Global chest pain score | Through study completion, an average of 1 year
  Will be evaluated by the Global chest pain score at the time of discharge from recovery area using a Visual Analog Scale 0-100 and represents the pain experienced by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Horiana Grosu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org